CLINICAL TRIAL: NCT02503176
Title: An Extension Study of KCT-0809 in Dry Eye Patients With Sjögren's Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinuation of the development
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KCT1302
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Dry Eye With Sjögren's Syndrome
Keywords: Dry eye syndromes; Corneal diseases; Conjunctival diseases
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases; Conjunctival Diseases

ARMS (1):
- KCT-0809 (Experimental)
  Interventions: Drug: KCT-0809 ophthalmic solution

INTERVENTIONS:
Drug: KCT-0809 ophthalmic solution

SUMMARY:
The purpose of this study is to evaluate of the long-term safety and efficacy of KCT-0809 in dry eye patients with Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye patients with Sjögren's syndrome finished KCT1301 study

Exclusion Criteria:

* Patients with poor adherence to medication of study drug in KCT1301 study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Incidences of adverse events | 52 weeks

SECONDARY OUTCOMES:
Score of the corneal staining | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan